CLINICAL TRIAL: NCT06258460
Title: Evaluating the Effectiveness of Multimodal Psychotherapy Training Program for Medical Students in China: Study Protocol for a Randomized Controlled Trial
Brief Title: Multimodal Psychotherapy Training for Chinese Medical Students
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sir Run Run Shaw Hospital (Other)
Responsible Party: Principal Investigator, Yanhui Liao, Attending Psychiatrist, Sir Run Run Shaw Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2024-0066
Record Dates: First submitted 2024-02-06; First posted 2024-02-14 (Actual); Last update posted 2024-02-20 (Actual); Status verified 2024-02

CONDITIONS: Mental Illness
Keywords: Multimodal teaching; psychotherapy training; Chinese medical students; randomized controlled trial
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Intervention Model Description: This study will be a two-arm randomized controlled trial (RCT). The intervention group will receive a two-day multimodal-based intensive educational intervention with 8 weeks follow-up (supervision based online teaching). The wait-list control group will not receive the intervention until the end of the study. Both groups will be followed up to 8 weeks.
Who Masked: Outcomes Assessor
Masking Description: Data will be blinded to intervention assignment by the trial statistician using R software
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the two-day psychotherapy training program with 8-week follow-ups intervention group (Experimental): All participants from the intervention group will receive the two-day psychotherapy training program. They will receive a hard copy booklet of the psychotherapy training program at recruitment. In addition, supervision-based group meeting will be hold at week 1, 2, 4, and 8 during follow-ups, and each meeting will be lasted for approximately two hours. At each follow-up meeting, the teachers, including psychotherapists and psychiatrists, will be prepared to answer any psychotherapy related questions, encourage them to practice psychological interventions, and provide more information for participants' clinical application of psychotherapy.
  Interventions: Other: psychotherapy training program intervention
- the wail-list control group (Placebo Comparator): After consent is given, participants who are allocated to the wail-list control group will receive a message encouraging them to complete all questionnaires from baseline to the last follow-up at 8 weeks. They will receive messages via WeChat to thank them for being in the study and reminding them of the time until the completion of the study at 8 weeks follow-up. They will receive a digital booklet of the psychotherapy training program via the WeChat individual messaging platform at recruitment, or a hard copy on request. After the trial ends, participants in the control arm will be able to receive the psychotherapy training program for free.
  Interventions: Other: the wail-list control intervention

INTERVENTIONS:
Other: psychotherapy training program intervention — The intervention group will receive a two-day multimodal-based intensive educational intervention of CBT with 8 weeks follow-up (supervision based online teaching).
  Arms: the two-day psychotherapy training program with 8-week follow-ups intervention group
Other: the wail-list control intervention — The wail-list control group will receive a message encouraging them to complete all questionnaires from baseline to the last follow-up at 8 weeks.
  Arms: the wail-list control group

SUMMARY:
Providing evidence-based, well-designed psychotherapy teaching to train them to get a basic understanding of psychotherapy and to gain required skills for clinical practice would be fundamental to medical students, residency. This study will be a two-arm randomized controlled trial (RCT) to evaluate the effectiveness of multimodal psychotherapy training program for medical students in China.

DETAILED DESCRIPTION:
Background and aims: Providing evidence-based, well-designed psychotherapy teaching for medical students and residents is urgently needed. The aim of this project is to measure the effectiveness of a newly multimodal psychotherapy teaching program for medical students and residents in China.

Design: This study will be a two-arm randomized controlled trial (RCT). The intervention group will receive a two-day multimodal-based intensive educational intervention with 8 weeks follow-up (supervision based online teaching). The wait-list control group will not receive the intervention until the end of the study. Both groups will be followed up to 8 weeks.

Setting: This trial will be conduct at the Sir Run Run Shaw Hospital.

Participants: This study aims to recruit about 160 medical students and residents, with approximately 80 in each group.

Measurements: The primary outcome measure is the changes of the Facilitative Interpersonal Skills task (FIS) scores. Secondary outcome measures include: training program acceptability; trainees' psychotherapy knowledge; utilization of psychotherapy; and self-reported self-efficacy and self-reported motivation for psychotherapy.

Comments: If this CBT-based brief and short-term psychotherapy skill training program is proven effective, the mental health impact of its expansion nation-wide could be enormous.

ELIGIBILITY:
Inclusion Criteria:

1. Medical student, residents, health care providers
2. 18 years of age or older
3. Expressing an interest in psychotherapy
4. Willingness to received randomization
5. Willing to provide informed consent to participate in the study

Exclusion Criteria:

1. Not health care providers
2. Below 18 years old
3. Unwilling to be randomized
4. Unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2014-02-01 (Actual); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-04-15 (Estimated)

PRIMARY OUTCOMES:
Facilitative Interpersonal Skills task (FIS) | 8 weeks
  FIS has eight dimensions: 1) verbal fluency, 2) hope and positive expectations, 3) persuasiveness; 4) emotional expression; 5) warmth, acceptance and understanding; 6) empathy; 7) alliance-bond capacity; and 8) alliance rupture-repair responsiveness. The items are rated on a 5-point Likert scale ranging from 1 (i.e., skill deficit) to 5 (i.e., optimal presence of skill), with high inter-rater agreement and excellent internal consistency. Research indicates that FIS is reliable measure to evaluate performance and psychotherapeutic outcomes in training and assessing therapists, high FIS indicate superior outcomes and better therapeutic processes. It measures therapists' demonstrated ability to convey psychotherapy's common factors, such as hopefulness, warmth, persuasiveness, and emotional engagement.

SECONDARY OUTCOMES:
Training program acceptability | 2 days
  program acceptability will be measured for participants from the intervention group by questions for assessing program acceptability
Trainees' psychotherapy knowledge | 8 weeks
  Knowledge about psychotherapy before and after 8 weeks will be on a 5-point scale
Utilization of psychotherapy | 8 weeks
  the utilization rate of psychotherapy interventions for patients during 8 weeks follow-up will be measured.
Self-reported self-efficacy | 8 weeks
  the self-efficacy will be measured by the visual analog scale (VAS) on a 10-cm line that represents a continuum between "no self-efficacy" and "the strongest self-efficacy."
Self-reported motivation | 8 weeks
  the motivation will be measured by the visual analog scale (VAS) on a 10-cm line that represents a continuum between "no motivation" and "the strongest motivation."

CONTACTS AND LOCATIONS:
Overall Officials: Tang Jinsong, MD, Study Director — Sir Run Run Shaw Hospital
Locations (1):
- Yanhui Liao, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
This study data will be shared with other researchers by requirement.

REFERENCES:
- [Derived] Ding Y, Pei T, Peng P, Yao J, Tang J, Liao Y. Attitudes and knowledge for CBT-based psychotherapy among medical students and residents in China: a survey study. BMC Med Educ. 2025 Jan 15;25(1):68. doi: 10.1186/s12909-025-06641-w. PMID 39815284
- [Derived] Pei T, Ding Y, Tang J, Liao Y. Evaluating the Effectiveness of a Multimodal Psychotherapy Training Program for Medical Students in China: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2025 Jan 3;14:e58037. doi: 10.2196/58037. PMID 39752191